CLINICAL TRIAL: NCT01486004
Title: A Phase-I, Open-label Trial in Healthy Female Subjects to Investigate the Effect of TMC435 at Steady-state on the Steady-state Pharmacokinetics of Ethinylestradiol and Norethindrone
Brief Title: A Study in Healthy Female Participants Investigating the Effect of TMC435 on the Pharmacokinetics of the Synthetic Hormones of the Oral Contraceptive Ovysmen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100683; TMC435-TiDP16-C124 (Other: Tibotec Pharmaceuticals); 2011-003022-26 (EudraCT Number)
Record Dates: First submitted 2011-10-21; First posted 2011-12-06 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Virus; TMC435; TMC435-TiDP16-C124; TMC435-C124; HCV; Hepatitis C; Hep C; Healthy participants
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): 35 µg ethinylestradiol and 1 mg norethindrone once daily for first 21 days in each OC cycle (2 OC cycles in total) + 150 mg capsule once daily for 10 days (Day12 till and including Day21) in 2nd OC cycle
  Interventions: Drug: TMC435; Drug: Ovysmen

INTERVENTIONS:
Drug: TMC435 — Type = exact number, unit = mg, number = 150, form = capsule, route = oral use. Capsule is taken once daily for 10 days (Day12 till and including Day21) in 2nd OC cycle.
Drug: Ovysmen — Type = exact number, unit = mg, number = 35µg/1mg, form = tablet, route = oral use. 35 µg ethinylestradiol and 1 mg norethindrone once daily for first 21 days in each OC cycle (2 OC cycles in total)

SUMMARY:
The purpose of this study is to investigate the effect of steady-state concentrations of TMC435 (administered once a day) on the steady-state pharmacokinetics of ethinylestradiol and norethindrone (administered once a day) and on the levels of progesterone, luteinizing hormone and follicle-stimulating hormone, in healthy female participants. Ethinlyestradiol and norethindrone are synthetic hormones, which constitute the oral contraceptive Ovysmen. Also the short-term safety and tolerability of the co-administration of TMC435 and Ovysmen will be studied. Steady-state is a term that means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. TMC435 is being investigated for the treatment of chronic hepatitis C virus (HCV) infection. Pharmacokinetics (PK) means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body. A contraceptive is a method that prevents pregnancy.

DETAILED DESCRIPTION:
This is a Phase I, open-label (both participant and investigator know the name of the medication given at a certain moment) trial in 18 healthy female participants to investigate the effect of TMC435 at steady-state on the steady-state pharmacokinetics of ethinlyestradiol and norethindrone. Ethinylestradiol (35 µg) and norethindrone (1.0 mg) are the components of Ovysmen, which is a widely used oral contraceptive (OC). All subjects will receive OC therapy for 2 complete OC cycles. During the first cycle, participants will receive Ovysmen alone, once daily, for the first 21 days. An OC- free period is respected from Day22 till and including Day28. During the second OC cycle, participants will receive again Ovysmen once daily during the first 21 days plus TMC435 150 mg once daily as of Day12 till and including Day21. Next, a OC-free period from Day22 till and including Day28 is established. Full 24-hour PK profiles of ethinylestradiol and norethindrone will be determined at the last day of OC treatment of the first OC cycle (i.e. on Day21) and on the last day of OC treatment of the second OC cycle (i.e. Day21). Full 24-hour PK profile of TMC435 will be determined on Day21 of second OC cycle. Pharmacodynamic (how the body reacts on the drug) assessments of serum levels of progesterone, luteinizing hormone and follicle-stimulating hormone (these hormones are involved in ovulation and in preparation of the womb for a pregnancy) will be done on Day1, 19, 20 and 21 of both OC cycles. Safety and tolerability will be assessed during the study period and during follow up. Blood and urine safety samples, electrocardiogram (ECG) and vital signs (blood pressure and heart rate) will be taken at screening, Day1, Day21 and Day22 of each OC cycle, and at the follow-up visit about 5 to 7 days after last TMC435 intake. A physical examination will be performed at screening, Day1 and Day20 of each OC cycle, and at the follow-up visit about 5 to 7 days after last TMC435 intake. Participants are admitted to the unit on Day20 in the morning and are discharged on Day22, for both OC cycles.

ELIGIBILITY:
Inclusion Criteria:

* Participants must practicing a highly effective method of birth control before entry and agree to continue to use the same method throughout the study and for at least 30 days after last administration of study drug
* non-smoker for a least 3 months prior to screening

Exclusion Criteria:

* Women who are pregnant, breastfeeding, pre-menopausal or post-menopausal
* A positive Human Immunodeficiency Virus (HIV)-1 or HIV-2 test at screening
* A positive Hepatitis A, B and C test at screening
* A clinical significant abnormal finding in the gynaecological examination

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in the steady-state plasma PK of ethinylestradiol following co-administration with TMC435 | Measured on Day19 till and including Day22 of 2nd OC cycle. Reference is Day19 till and including Day22 of 1st OC cycle.
  PK characteristics of ethinylestradiol and norethindrone are determined based on their respective plasma levels at one time point (Day19, 20 and 22) and at 10 time points (Day22). Standard PK parameters such as C0h, Cmin, Cmax, Tmax, AUC24h etc. will be determined.
Change in the steady-state plasma PK of norethindrone following co-administration with TMC435 | Measured on Day19 till and including Day22 of 2nd OC cycle. Reference is Day19 till and including Day22 of 1st OC cycle.
  PK characteristics of ethinylestradiol and norethindrone are determined based on their respective plasma levels at one time point (Day19, 20 and 22) and at 10 time points (Day22). Standard PK parameters such as C0h, Cmin, Cmax, Tmax, AUC24h etc. will be determined.

SECONDARY OUTCOMES:
Change in the plasma levels of progesterone following co-administration of Ovysmen and TMC435. | Measured on Day1, 19, 20 and 21 of 2nd OC cycle. Reference is Day1, 19, 20 and 21 of 1st OC cycle.
  Plasma levels of progesterone.
Number of participants (%) with adverse events as a measure of safety and tolerability when combining TMC435 (150 mg, q.d.) with Ovysmen (35 µg ethinylestradiol + 1 mg norethindrone, q.d.) | Day of Screening + 21 days between screening and Day1 of first OC cycle + 28 days of first OC cycle + 28 days of second OC cycle
Change in the plasma levels of luteinizing hormone following co-administration of Ovysmen and TMC435. | Measured on Day1, 19, 20 and 21 of 2nd OC cycle. Reference is Day1, 19, 20 and 21 of 1st OC cycle.
  Plasma levels of luteinizing hormone.
Change in the plasma levels of follicle-stimulating hormone following co-administration of Ovysmen and TMC435. | Measured on Day1, 19, 20 and 21 of 2nd OC cycle. Reference is Day1, 19, 20 and 21 of 1st OC cycle.
  Plasma levels of follicle-stimulating hormone.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (1):
- Merksem, Belgium